CLINICAL TRIAL: NCT06739330
Title: Thyroid Dysfunction and Its Association With Metabolic Dysfunction-Associated Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shimaa Abdelmounem Meshaal, Lecturer of Tropical Medicine and Infectious Diseases, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR929/11/24
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Dysfunction; Metabolic Dysfunction-Associated Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with metabolic dysfunction-associated fatty liver disease (MAFLD)
  Interventions: Device: Fibroscan
- Control group: Healthy control patients
  Interventions: Device: Fibroscan

INTERVENTIONS:
Device: Fibroscan — Fibroscan will be used to assess the stages of fibrosis and steatosis using Dimensional ultrasound TE (transient elastography). Dimensional ultrasound TE (transient elastography) will be used for staging liver fibrosis and steatosis by measuring the velocity of a low frequency (50 Hz) elastic shear wave propagating through the liver.

SUMMARY:
This study aims to evaluate the prevalence of thyroid dysfunction and its association with metabolic dysfunction-associated fatty liver disease.

DETAILED DESCRIPTION:
One of the most common causes of chronic liver diseases worldwide is metabolic dysfunction-associated fatty liver disease (MAFLD), which affects about 30% of adults. Thyroid hormones are critical in maintaining metabolic homeostasis throughout life and are intimately linked to the liver.

Dysfunctions of the thyroid gland have been implicated as one of the most important risk factors of MAFLD due to its important role in the hepatic synthesis of fatty acid and cholesterol. Maintaining liver metabolism requires thyroid function to be normal, while thyroid disorders may lead to liver disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients with metabolic dysfunction-associated fatty liver disease (MAFLD).

Exclusion Criteria:

* History of thyroid disease or treatment (e.g., thyroid nodules, thyroid cancer, hypothyroidism, and hyperthyroidism).
* Patients with alcoholic liver disease take more than 40g of alcohol (or four units) per day.
* Viral hepatitis.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional case-control study will be carried out on 150 patients with metabolic dysfunction-associated fatty liver disease (MAFLD) at Tanta University Hospitals for a period from October 2024 to April 2025 after approval from the Institutional Ethical Committee.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Level of free triiodothyronine (FT3) | After the sample is taken (up to 5 minutes)
  Free triiodothyronine (FT3) will be measured using chemiluminescent immunoassay analysis.

SECONDARY OUTCOMES:
Level of free thyroxine (FT4) | After the sample is taken (up to 5 minutes)
  Free thyroxine (FT4) will be measured using chemiluminescent immunoassay analysis.
Level of thyroid stimulating hormone | After the sample is taken (up to 5 minutes)
  Thyroid stimulating hormone will be measured using chemiluminescent immunoassay analysis.
Relation between gender and thyroid function | After the sample is taken (up to 5 minutes)
  Relation between gender and thyroid function will be assessed.
Correlation between metabolic data and thyroid function tests | After the sample is taken (up to 5 minutes)
  Correlation between metabolic data and thyroid function tests will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.